CLINICAL TRIAL: NCT06014580
Title: Molecular and Epidemiological Characteristics of Endometrial Cancer in Brazil
Acronym: MADONNA
Status: Active, not recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 0521
Record Dates: First submitted 2023-06-15; First posted 2023-08-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with endometrial cancer: Patients diagnosed with endometrial cancer between January 2016 and December 2019 at participating sites will be included.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study; patients will not be exposed to clinical interventions different from those belonging to the standard of care.

SUMMARY:
An evaluation of the molecular and epidemiological aspects of endometrial cancer in Brazil is necessary to understand the high frequency of advanced disease. A better understanding of the current situation will generate essential data for the future development of national or international cooperative programs that aim to improve outcomes in these patients and generate additional knowledge for much-needed clinical trials in this population.

DETAILED DESCRIPTION:
This is a retrospective observational cohort study. In this study, we will include patients diagnosed with endometrium cancer from January 2016 to December 2019 in participating sites and collect data on demographics, clinicopathological characteristics, treatment patterns, and outcomes. Data will be collected from medical records in selected centers that comprise different regions of Brazil.

The patient data sources will be the medical records of the patients. Patients will continue to receive treatment and clinical evaluations for endometrial cancer according to what is determined by their medical team, according to the usual standards of treatment and clinical practice of each center. To minimize patient selection bias, physicians should invite all consecutive eligible patients.

This study also provides for the collection and archiving of tumor tissue material. The samples will be tested to characterize the molecular subtype of endometrial cancer and will be sequentially stored in a biorepository to enable future translational studies, according to national regulations.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years
* Histological diagnosis of endometrial carcinoma.
* Diagnosis of endometrial cancer between January 2016 and December 2019.
* FIGO (International Federation of Gynecology and Obstetrics, 2018) Stage I - IV.
* Site and investigator with access to a medical record chart from which data can be abstracted.
* Presence of a sample of tumor tissue (primary tumor or metastasis) available for biomarker testing.

Exclusion Criteria:

* Noninvasive endometrial cancer.
* Patients with a history of concurrent or previously treated non-endometrial malignancies except for appropriately treated 1) non -metastatic non-melanoma skin cancer and/or 2) non-metastatic low-grade thyroid tumors and/or 3) in situ carcinomas, including cervix, colon, and skin.
* Nonepithelial histology (leiomyosarcoma, adenosarcoma, endometrial stromal sarcoma, undifferentiated sarcoma, or other mesenchymal tumors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with endometrial cancer between January 2016 and December 2019 at participating research sites.
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiological Characteristics of the Brazilian Population with Endometrial Cancer | At the time of diagnosis.
  This measure encompasses key epidemiological factors of the Brazilian population diagnosed with endometrial cancer, including age distribution, racial and ethnic demographics, geographic regions, and relevant comorbidities. These details will provide insights into the demographic makeup of the study population.
Molecular Profile Analysis of Endometrial Cancer Cases | Throughout the study period, an average of 36 month.
  This measure focuses on analyzing the molecular profile of endometrial cancer cases in the Brazilian population. It includes information about specific genetic mutations, biomarkers, and molecular subtypes that are relevant to endometrial cancer. Understanding the molecular landscape can contribute to insights into disease progression and potential targeted therapies.
Treatment Patterns for Endometrial Cancer in Brazil | From diagnosis to completion of treatment, between January 2016 and December 2019.
  This measure examines the treatment patterns employed for endometrial cancer within the Brazilian population. It includes details about types of treatments received, such as surgery, chemotherapy, radiation therapy, and hormonal therapy. Additionally, it explores the utilization of targeted therapies or immunotherapies.
Endometrial Cancer Outcomes in the Brazilian Population | From diagnosis to the end of the study follow-up period, an average of 36 months.
  This measure assesses the outcomes of endometrial cancer cases in the Brazilian population. It includes survival rates, disease recurrence rates, response to treatment, and overall disease progression. By evaluating these outcomes, a comprehensive understanding of the disease's impact on the population can be achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia Cristina de Melo, Principal Investigator — Latin American Cooperative Oncology Group
Locations (7):
- Brazil (7):
  - ICC - Instituto do Câncer do Ceará, Fortaleza, Ceará
  - Hospital Evangélico de Cachoeiro de Itapemirim - Centro de Pesquisas Clínicas em Oncologia (CPCO), Cachoeiro de Itapemirim, Espírito Santo
  - Santa Casa de Misericórdia de Feira de Santana, Feira de Santana, Estado de Bahia
  - Clinica Prognóstica - Centro de Pesquisa Clínica Onconeo, Campo Grande, Mato Grosso do Sul
  - Instituto do Câncer Brasil - Unidade Três Lagoas, Três Lagoas, Mato Grosso do Sul
  - UOPECCAN - Hospital do Câncer de Cascavel, Cascavel, Santa Catarina
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Undecided